CLINICAL TRIAL: NCT02815215
Title: A Retrospective Multicenter Analysis on Treatment of Congenital Idiopathic Clubfoot With Minimally Invasive Carroll's Technique
Brief Title: Efficacy Analysis of Minimally Invasive Carroll's Technique in Treatment of Congenital Idiopathic Clubfoot
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LiMing (Other)
Collaborators: Hunan Children's Hospital (Other Government); Shenzhen Children's Hospital (Other Government); Guangzhou Women and Children's Medical Center (Other)
Responsible Party: Sponsor-Investigator, LiMing, Chief of Pediatric Orthopedics, Children's Hospital of Chongqing Medical University
Organization: Children's Hospital of Chongqing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHChongqingMU
Record Dates: First submitted 2016-06-21; First posted 2016-06-28 (Estimated); Last update posted 2016-06-28 (Estimated); Status verified 2016-06

CONDITIONS: Congenital Clubfoot
Keywords: congenital clubfoot
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention group (Experimental): Minimally Invasive Carroll's Technique
  Interventions: Procedure: Minimally Invasive Carroll's Technique
- Control group (Active Comparator): Ponseti method
  Interventions: Procedure: Ponseti method

INTERVENTIONS:
Procedure: Minimally Invasive Carroll's Technique — Patient will be treated with minimally invasive Carroll's technique by 3 small incisions in the heel, in the medial side of the foot and in the planta pedis, respectively. Long-leg plaster cast fixation was applied for 6-8 weeks
  Arms: Intervention group
Procedure: Ponseti method — As a control, Patient will be treated with classical Ponseti method, including multiple steps: manipulative correction, continuous plaster, achilles tendon cutting, fixation.
  Arms: Control group

SUMMARY:
Congenital clubfoot(CCF) is a kind of common congenital foot deformities in children. Though Ponseti method can cure most of the CCF patients, there are still part of patients can not get satisfactory recovery, especially those children classified as Dimeglio grade Ⅲ and Ⅳ. Carroll's technique is considered to be an ideal method of surgical treatment. But the postoperative scar is relatively large, and accordingly the postoperative complications is still common. Based on the clinical practice of the investigator's group, a modification of Carroll's technique, minimally invasive Carroll's technique, was applied. For the Dimeglio grade Ⅲ and Ⅳ CCF, the postoperative excellent and good rate was over 90%. Therefore, the investigator conducted a multicenter randomized controlled trial on treatment of congenital idiopathic clubfoot with minimally invasive Carroll's technique.

ELIGIBILITY:
Inclusion Criteria:

* First diagnosed congenital idiopathic clubfoot cases classified as Dimeglio grade Ⅲ and Ⅳ

Exclusion Criteria:

* Age≤28 days, and Age>4 years.
* Accompanied by serious diseases of other organs.
* Children with inherited metabolic disease and connective tissue disease.
* Clubfoot caused by trauma, cerebral palsy, congenital multiple joint contracture, polio, spina bifida occulta, and clubfoot derived from spinal cord disease.

Ages: 28 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Dimeglio classification system | 0 month(before treatment); 3rd month, 1st year, 3rd year(after treatment)
  evaluate the grade before and after treatment

SECONDARY OUTCOMES:
Pirani scoring system | 0 month(before treatment); 3rd month, 1st year, 3rd year(after treatment)
  evaluate the grade before and after treatment

OTHER OUTCOMES:
talocalcaneal angle measurement | 0 month(before treatment); 3rd month, 1st year, 3rd year(after treatment)
  evaluate the grade before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ming Li, master, Principal Investigator — Children's Hospital of Chongqing Medical University
Locations (1):
- Children's Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Carroll NC. Clubfoot in the twentieth century: where we were and where we may be going in the twenty-first century. J Pediatr Orthop B. 2012 Jan;21(1):1-6. doi: 10.1097/BPB.0b013e32834a99f2. PMID 21946867